CLINICAL TRIAL: NCT01363856
Title: Center for Stroke Research Berlin (CSB) Prospective Stroke Cohort
Acronym: CSB_PROSCIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Klinikum der Universitaet Muenchen, Grosshadern (Other)
Responsible Party: Matthias Endres, MD, Center for Stroke Research Berlin
Other Study IDs: CSB_PROSCIS_01
Record Dates: First submitted 2011-05-31; First posted 2011-06-02 (Estimated); Last update posted 2011-06-02 (Estimated); Status verified 2011-05

CONDITIONS: Stroke
Keywords: first ever stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples with DNA whole blood, serum, RNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- First ever acute stroke: Patients over 18 years and without prior stroke according to WHO criteria, displaying an ischemic stroke, onset within the last 7 days, language German

SUMMARY:
The primary aim of the study is to derive and validate risk scores for vascular endpoints (recurrent stroke, myocardial infarction, and other complications of stroke) and for death following an incident stroke. For this purpose patients with an incident stroke will be followed for 36 months with additional assessments at 12, 24 and 36 months.

DETAILED DESCRIPTION:
Risk of vascular disease including stroke, myocardial infarction, and vascular death is high after stroke but there are only few prognostic models for long term risk up to 3 years. About 850 patients with an incident stroke will be followed for 3 years with assessments at baseline and at 3, 12, 24, and 36 months. Factors that have already been reported to be significant predictors of vascular diseases in previous studies as well as new biomarkers (e.g. neuroimaging, blood based biomarkers) identified in this cohort will be considered. The improvement of discrimination including these new variables in the models will be investigated. Several measures of improving predictive properties (e.g. calibration, discrimination, net reclassification) will be used to compare predictive models with different complexity. The model will be validated using the bootstrap method (internal validation) and an independent external sample in cooperation with the Institute for Stroke and Dementia Research, Munich.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Language: German
* First ever stroke including ischemic stroke, primary intracranial hemorrhage and cerebral venous sinus thrombosis that occurred with stroke onset in the last 7 days
* Written informed consent by patient prior to study participation
* Willingness to participate in follow-up

Exclusion Criteria:

* Prior stroke (definition according to WHO definition)
* Patients presenting brain tumour or brain metastasis
* Participation in an intervention- / AMG-study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to a specialized stroke service because of an acute stroke
Sampling Method: Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2010-02; Primary Completion 2013-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Combined vascular endpoint composed of stroke, myocardial infarction, and vascular death | 36 months
  This evaluation will be based on a structured interview with the patient. In case of positive screening more information will be obtained by hospital or physician.

SECONDARY OUTCOMES:
Combined vascular endpoint composed of stroke, myocardial infarction, and vascular death | 24 months
  This evaluation will be based on a structured interview with the patient. In case of positive screening more information will be obtained by hospital or physician. In case of death of the patient, evaluation will be based on data from the registry office
Combined vascular endpoint composed of stroke, myocardial infarction, and vascular death | 12 months
  This evaluation will be based on a structured interview with the patient. In case of positive screening more information will be obtained by hospital or physician. In case of death of the patient, evaluation will be based on data from the registry office
Course of cognitive function | 36 months
  This evaluation will be based on a structured interview with the patient. In case of positive screening more information will be obtained by the physician
Course of depression | 36 months
  This evaluation will be based on a structured interview with the patient. In case of positive screening more information will be obtained by the physician

CONTACTS AND LOCATIONS:
Overall Officials: Peter U Heuschmann, MD MPH, Principal Investigator — Center for Stroke Research Berlin, Charité Campus Mitte
Locations (2):
- Germany (2):
  - Center for Stroke Research Berlin, Charité Universitätsmedizin Berlin, Berlin, State of Berlin
  - Interdisciplinary Stroke Center Munich, Klinikum der Universität München, Campus Großhadern, Munich

REFERENCES:
- [Derived] Giesers NK, Schaeff V, Gertz K, Endres M, Liman TG. Associations of Soluble Inflammatory and Endothelial Activation Biomarkers with Cognitive Function Over Three Years After Ischemic Stroke-PROSCIS-B. Transl Stroke Res. 2025 Dec;16(6):2249-2257. doi: 10.1007/s12975-025-01388-4. Epub 2025 Oct 8. PMID 41057606
- [Derived] Rios AS, Temuulen U, Khalil AA, Villringer K, Ali HF, Akdeniz A, Grittner U, Becher M, Rackoll T, Nave AH, Sperber PS, Liman TG, Otte C, Endres M, Kufner A. Lesion-Network Mapping of Poststroke Depressive Symptoms: Evidence From Two Prospective Ischemic Stroke Cohorts. Stroke. 2025 Sep;56(9):2527-2539. doi: 10.1161/STROKEAHA.125.051858. Epub 2025 Jul 7. PMID 40620229
- [Derived] Liman TG, Siegerink B, Piper S, Catar R, Moll G, Riemekasten G, Heidecke H, Heuschmann PU, Elkind MSV, Dragun D, Endres M. Vasoregulatory Autoantibodies and Clinical Outcome After Ischemic Stroke-PROSCIS-B. J Am Heart Assoc. 2023 Dec 5;12(23):e032441. doi: 10.1161/JAHA.123.032441. Epub 2023 Nov 28. PMID 38014691
- [Derived] Schaeff VLK, Sperber PS, Piper SK, Giesers NK, Gertz K, Heuschmann PU, Endres M, Liman TG. Associations of C-reactive protein with depressive symptoms over time after mild to moderate ischemic stroke in the PROSCIS-B cohort. J Neurol. 2024 Feb;271(2):909-917. doi: 10.1007/s00415-023-12038-w. Epub 2023 Oct 18. PMID 37848651
- [Derived] Stillfried MRV, Sperber PS, Broersen LHA, Huo S, Piper SK, Heuschmann PU, Endres M, Siegerink B, Liman TG. Low ankle-brachial index and cognitive function after stroke-the PROSpective with Incident Stroke Berlin (PROSCIS-B). Front Neurol. 2022 Sep 28;13:963262. doi: 10.3389/fneur.2022.963262. eCollection 2022. PMID 36247749
- [Derived] Scheitz JF, Lim J, Broersen LHA, Ganeshan R, Huo S, Sperber PS, Piper SK, Heuschmann PU, Audebert HJ, Nolte CH, Siegerink B, Endres M, Liman TG. High-Sensitivity Cardiac Troponin T and Recurrent Vascular Events After First Ischemic Stroke. J Am Heart Assoc. 2021 May 18;10(10):e018326. doi: 10.1161/JAHA.120.018326. Epub 2021 May 13. PMID 33982599
- [Derived] Huo S, Krankel N, Nave AH, Sperber PS, Rohmann JL, Piper SK, Heuschmann PU, Landmesser U, Endres M, Siegerink B, Liman TG. Endothelial and Leukocyte-Derived Microvesicles and Cardiovascular Risk After Stroke: PROSCIS-B. Neurology. 2021 Feb 9;96(6):e937-e946. doi: 10.1212/WNL.0000000000011223. Epub 2020 Nov 12. PMID 33184230
- [Derived] Broersen LHA, Siegerink B, Sperber PS, von Rennenberg R, Piper SK, Nolte CH, Heuschmann PU, Endres M, Scheitz JF, Liman TG. High-Sensitivity Cardiac Troponin T and Cognitive Function in Patients With Ischemic Stroke. Stroke. 2020 May;51(5):1604-1607. doi: 10.1161/STROKEAHA.119.028410. Epub 2020 Apr 13. PMID 32279621
- [Derived] Sperber PS, Siegerink B, Huo S, Rohmann JL, Piper SK, Pruss H, Heuschmann PU, Endres M, Liman TG. Serum Anti-NMDA (N-Methyl-D-Aspartate)-Receptor Antibodies and Long-Term Clinical Outcome After Stroke (PROSCIS-B). Stroke. 2019 Nov;50(11):3213-3219. doi: 10.1161/STROKEAHA.119.026100. Epub 2019 Sep 17. PMID 31526121
- [Derived] Liman TG, Zietemann V, Wiedmann S, Jungehuelsing GJ, Endres M, Wollenweber FA, Wellwood I, Dichgans M, Heuschmann PU. Prediction of vascular risk after stroke - protocol and pilot data of the Prospective Cohort with Incident Stroke (PROSCIS). Int J Stroke. 2013 Aug;8(6):484-90. doi: 10.1111/j.1747-4949.2012.00871.x. Epub 2012 Aug 29. PMID 22928669
- See also: Center for Stroke Research Berlin — http://www.strokecenter.de